CLINICAL TRIAL: NCT05300854
Title: Serratus Anterior Plane Block Versus Paravertebral Plane Block for Post Thoracotomy Pain Relief: A Comparative Study
Brief Title: Serratus Block Versus Paravertebral Block for Post Thoracotomy Pain Relief
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Eman Ibraheem Darweesh, lecturer of anesthesia and intensive care, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: soh-Med-22-2-23
Record Dates: First submitted 2022-03-19; First posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard anesthesia in addition to serratus plane block (Active Comparator): general anesthesia was given then ultrasound-guided serratus plane block
  Interventions: Procedure: Standard anesthesia in addition to serratus plane block
- Standard anesthesia in addition to para-vertebral block (Active Comparator): general anesthesia was given then ultrasound-guided para-vertebral block
  Interventions: Procedure: Standard anesthesia in addition to para-vertebral block

INTERVENTIONS:
Procedure: Standard anesthesia in addition to serratus plane block — a US-guided SPB was performed after induction of general anesthesia with the patient lying supine.
  Arms: Standard anesthesia in addition to serratus plane block
Procedure: Standard anesthesia in addition to para-vertebral block — Standard anesthesia in addition to para-vertebral block
  Arms: Standard anesthesia in addition to para-vertebral block

SUMMARY:
This double-blinded, randomized controlled study was done on 60 patients older than 18 years undergoing thoracotomy. Patients were allocated into two equal groups (30 patients each). Group S: Standard anesthesia in addition to SPB. II. Group P: Standard anesthesia in addition to PVB.

ELIGIBILITY:
Inclusion Criteria:

* patients more than 18 ys undergoing thoracotomy operation

Exclusion Criteria:

* morbid obesity (Body mass index > 40)
* impossibility of anatomical structures US identification in a satisfactory way
* opioids treatment before surgery or substance abuse,
* sepsis and/or infection at the puncture sites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
prevention of post-operative pain | 72 hours
  reduction of visual analogue score
reduction of analgesic requirement | 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No